CLINICAL TRIAL: NCT01630070
Title: A Prospective, Multi-center, Single Arm Study With a Nitinol Self-Expanding Paclitaxel-Eluting Stent in the Treatment of Atherosclerotic Tibial-peroneal Arteries
Brief Title: Single Arm Study With a Nitinol Self-Expanding Paclitaxel-Eluting Stent to Treat BTK Arteries
Acronym: PES-BTK-70
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-110629
Record Dates: First submitted 2012-06-18; First posted 2012-06-28 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Critical limb ischemia; Rest pain; Minor tissue loss; Below the knee
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self-expandable drug eluting stent (Experimental): Self-Expanding Paclitaxel-Eluting stent
  Interventions: Device: Self-expandable drug eluting stent

INTERVENTIONS:
Device: Self-expandable drug eluting stent — Self-Expanding Paclitaxel-Eluting stent
  Other Names: Self-Expanding Paclitaxel-Eluting stent

SUMMARY:
The objective of this clinical study is to evaluate the immediate and long-term (up to 12 month) safety and effectiveness of a Nitinol Self-Expanding Paclitaxel-Eluting stent for the treatment of patients with critical limb ischemia (i.e. rest pain or non-healing foot ulcers) due to the presence of arterial lesions in the below-the-knee arteries of maximally 50mm long.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with rest pain or minor tissue loss (Rutherford Clinical Category 4 or 5)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 12 months
* Patient is eligible for treatment with a Self-Expanding Paclitaxel-Eluting stent
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure
* Evidence at screening of ≥50% de novo lesion (or restenosis after previous PTA) in the infrapopliteal arteries, confirmed by angiography
* Reference vessel diameter visually estimated to be ≥3.0mm and ≤4.5mm
* Identifiable distal target vessel which upon completion of the intervention, is anticipated to provide reconstitution of blood flow to the foot.
* Guidewire successfully traversed lesion
* Length of target lesion is <50mm

Exclusion Criteria:

* Untreated flow-limiting inflow lesions
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Has had a previous peripheral bypass affecting the target limb
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Non-atherosclerothic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Patient has a contra-indication or known untreated allergy to anti-platelet therapy, anticoagulants, thrombolytic drugs or any other drug anticipated to be used
* Patient has hypersensitivity to contrast or device material that cannot be adequately pretreated
* Patient has known uncontrollable hypercoagulable condition, or refuses blood transfusion
* Life expectancy of less than 12 months
* Patient is currently participating in an investigational drug or another device study that may clinically interfere with the study endpoints
* Patient has other co-morbid condition(s) that in the judgment of the physician precludes safe percutaneous intervention
* Has end-stage renal disease defined as undergoing hemodialysis for kidney failure
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT)type II
* Treatment of ipsilateral non-study inflow lesions with other materials than regular guidewires, regular PTA balloons, bare metal stents and/or paclitaxel-coated stents
* Additional treatments of the study lesion requiring materials/procedures other than standard guidewires, regular PTA balloons and/or a Self-Expanding Paclitaxel-Eluting stent (e.g. thrombectomy, re-entry catheters, CTO-wires, cutting balloon, cryoballoon, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary patency | 6 months
  Primary patency rate at 6 months, defined by duplex ultrasound measurement of peak systolic velocity ratio ≤2.0 at the target lesion(s) with no clinically-driven reintervention within the treated segment, verified by Core Lab
Primary patency | 12 months
  Primary patency at 12 months, defined as absence of restenosis (≥50% stenosis) or occlusion within the originally treated lesion based on angiography, verified by Core Lab

SECONDARY OUTCOMES:
Technical success | procedure (day 0)
  Technical success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30% by visual assessment
Procedural success | Procedure (day 0)
  Procedural success, defined as the ability to achieve <30% final residual stenosis of the target lesion by visual estimation (angio) and the absence of any in-hospital Major Adverse Events (MAE, defined as clinically-driven target vessel revascularization, major unplanned amputation of the treated limb, and all-cause mortality)
MAE (Major Adverse Event) | 1, 6 and 12 months
  MAE at 1, 6 and 12 months
  Major Adverse Events (MAE) include (but are not limited to)
  * death
  * myocardial infarction
  * stroke
  * emergent surgical revascularization of the target vessel
  * repeat vascularization of the target vessel
  * major amputation
  * bleeding complication requiring transfusion
SAE (Serious Adverse Event) | discharge, 1, 6 and 12 months
  Other SAEs at discharge, 1, 6 and 12 months
  A Serious Adverse Event (SAE) is defined as an Adverse Event which:
  * results in death
  * is life-threatening
  * results in persistent or significant disability/incapacity
  * requires in-patient hospitalization or unduly prolonged hospitalization.
  * necessitates an intervention to prevent a permanent impairment of a body function or permanent damage to a body structure.
  * is a congenital abnormality/birth defect, a fetal distress or fetal death
  * results in malignancy
Improvement of Rutherford classification | 12 months
  Improvement in Rutherford Clinical Category at 12 months, defined as an improvement in clinical status indicated by a decrease of one or more in Rutherford Clinical Category at 12 months compared to baseline, that is attributable to the treated limb (in cases of bilateral disease)
Improvement in Ankle-Brachial Index | 12 months
  Improvement in Ankle-Brachial Index at 12 months, defined as an increase in the ankle-brachial index (ABI) at 1 year compared to baseline in subjects with compressible arteries and baseline ABI<0.9
Primary Patency | 1 and 12 months
  Primary patency rate at 1 and 12 months, defined by duplex ultrasound measurement of peak systolic velocity ratio ≤2.0 at the target lesion(s) with no clinically-driven reintervention within the treated segment
Secondary patency | 1, 6 and 12 months
  Secondary patency rate at 1, 6 and 12 months, defined by duplex ultrasound peak systolic velocity ratio ≤2.0 maintained by repeat percutaneous intervention
Limb salvage rate | Procedure, 1, 6 and 12 months
  Limb salvage rate, defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot
Target Lesion Revascularisation | Procedure (day 0), 1, 6 and 12 months
  Target lesion revascularization (TLR), defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius
Locations (5):
- Belgium (5):
  - Imelda Hospital, Bonheiden, Antwerp
  - UZA, Edegem, Antwerp
  - RZ Heilig-Hartziekenhuis, Tienen, Antwerp
  - OLV Ziekenhuis, Aalst, East-Flanders
  - AZ Sint-Blasius, Dendermonde, East-Flanders

REFERENCES:
- [Derived] Bosiers M, Callaert J, Keirse K, Hendriks JMH, Peeters P, Verbist J, Maene L, Beelen R, Deloose K. One-Year Outcomes of the Paclitaxel-Eluting, Self-Expanding Stentys Stent System in the Treatment of Infrapopliteal Lesions in Patients With Critical Limb Ischemia. J Endovasc Ther. 2017 Jun;24(3):311-316. doi: 10.1177/1526602817697319. Epub 2017 Mar 9. PMID 28351310